CLINICAL TRIAL: NCT03877731
Title: Role of Mitral Valve in the Obstruction of Left Ventricular Outflow Tract in Patients With Hypertrophic Cardiomyopathy
Brief Title: Mitral Valve in Hypertrophic Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCMP-MV151
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-03

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: hypertrophic cardiomyopathy, mitral valve, echocardiography
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- hypertrophic cariomyopathy, isolated septal myectomy (Active Comparator): Patients with hypertrophic obstructive cardiomyopathy who will undergo isolated septal myectomy
  Interventions: Procedure: isolated septal myectomy
- hypertrophic cariomyopathy, septal myectomy + edge-to-edge (Experimental): Patients with hypertrophic obstructive cardiomyopathy who will undergo septal myectomy and edge-to-edge mitral valve repair (O. Alfieri technique)
  Interventions: Procedure: septal myectomy + edge-to-edge mitral valve repair
- hypertrophic cariomyopathy, septal myectomy + sliding plasty (Experimental): Patients with hypertrophic obstructive cardiomyopathy who will undergo septal myectomy and posterior leaflet sliding plasty ( A. Carpentier technique)
  Interventions: Procedure: septal myectomy + posterior leaflet sliding plasty
- hypertrophic cariomyopathy, septal myectomy + chordae (Experimental): Patients with hypertrophic obstructive cardiomyopathy who will undergo septal myectomy and secondary chordae transection
  Interventions: Procedure: septal myectomy + secondary chordae transection
- Arterial hypertension + left ventricular hypertrophy (No Intervention): Patients with arterial hypertension with left ventricular hypertrophy whose mitral valve geometry and papillary muscles' function will be compared to those of the patients with hypertrophic cardiomyopathy
- Control (No Intervention): Patients without structural heart disease whose mitral valve geometry and papillary muscles' function will be compared to those of the patients with hypertrophic cardiomyopathy

INTERVENTIONS:
Procedure: isolated septal myectomy
  Arms: hypertrophic cariomyopathy, isolated septal myectomy
Procedure: septal myectomy + edge-to-edge mitral valve repair
  Arms: hypertrophic cariomyopathy, septal myectomy + edge-to-edge
Procedure: septal myectomy + posterior leaflet sliding plasty
  Arms: hypertrophic cariomyopathy, septal myectomy + sliding plasty
Procedure: septal myectomy + secondary chordae transection
  Arms: hypertrophic cariomyopathy, septal myectomy + chordae

SUMMARY:
The purpose of the study is to assess the role of mitral valve apparatus in the development of outflow tract obstruction in patients with hypertrophic cardiomyopathy and to identify the best surgical treatment modality to relieve outflow tract obstruction in such patients

DETAILED DESCRIPTION:
It is well-known that mitral valve plays an important role in the development of left ventricular outflow tract obstruction in patients with hypertrophic cardiomyopathy. In order to further investigate this phenomenon, the following study aims to compare mitral valve geometry indices, as assessed by transthoracic echocardiography, two- and three-dimentional transesophageal echocardiography and mitral valve quantification analysis, and papillary musles' function, as assessed by 2D speckle tracking imaging, in patients with hypertrophic obstructive cardiomyopathy, patients with arterial hypertension and left ventricular hypertrophy and people without structural heart disease. This will provide information on the geometric characteristics of mitral valve that predispose to the development of obstruction. Futhermore, patients with hypertrophic obstructive cardiomyopathy that are eligible for the surgical relief of obstruction will be randomised into four groups according to the modality of intervention. These groups are as follows: 1) isolated extended septal myectomy; 2) extended septal myectomy + edge to edge mitral valve repair; 3) extended septal myectomy + posterior lealfet sliding plasty; 4) extended septal myectomy + secondary chordae transection. After surgery, said indices will be reassessed and the degree of outflow tract obstruction relief noted, in order to elicit which geometrical changes are produced by each type of intervention. Patients will be followed long-term, up to 5 years, in order to define whether the addition of the intervention on mitral valve helps abolish the residual gradient more effectively, and whether it translates into any survival benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed informed consent to participate in the study
* For patients with hypertrophic cardiomyopathy only: resting or latent peak left ventricular outflow tract gradient >50 mmHg, NYHA class III-IV
* For patients with arterial hypertension only: hystory of arterial pressure increase >140/90 mmHg, increased left vantricular wall thickness (>10 mm) and myocardial mass indexed to BSA (>95 g/m2 for women and >115 g/m2 for men), as assessed by 2D transthoracic echocardiography

Exclusion Criteria:

* Age < 18 years
* Persistent form of atrial fibrillation
* Intrinsic mitral or aortic valve disease
* Coronary artery disease
* Reduced left ventricular ejection fraction
* For control group only: presence of any structural heart disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  patients' survival without hospital admissions due to the recurring sympthoms

SECONDARY OUTCOMES:
Residual left vetricular outflow tract gradient | 5 years
  left ventricular outflow tract gradient measured by continuous doppler from 5-chamber apical view
Mitral regurgitation | 5 years
  degree of mitral regurgitation assessed by color doppler, regurgitant volume measured using PISA method
Papillary muscles' funcion | 5 years
  papillary muscles' strain and strain rate assessed by 2D speckle tracking imaging
Mitral valve geometry | 10 days
  indices of mitral valve geometry assessed by 2D transthoracic and transesophageal echocardiography and mitral valve quantification analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pavlyukova, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk NRMC
Locations (1):
- Cardiology research institute, National Research Medical Center of the Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No